CLINICAL TRIAL: NCT04451915
Title: Late Versus Early Management of Gestational Diabetes Mellitus: a Non Inferiority Randomized Multicenter Trial
Brief Title: Early Gestational Diabetes Mellitus
Acronym: LEMA_GDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017_76; 2018-A00794-51 (Other: ID-RCB number, ANSM); PHRC-17-008 (Other: PHRC number, DGOS)
Record Dates: First submitted 2020-06-22; First posted 2020-06-30 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Gestational Diabetes
Keywords: Early gestational diabetes; pregnancy; fasting plasma glucose; diagnosis; prognosis
MeSH Terms: conditions — Diabetes, Gestational; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early management GDM group (Experimental): defined as no intervention until GDM screening at 24-28 weeks' gestation. If there is a diagnosis of GDM at 24-28 according to the IADPSG criteria), intensive metabolic treatment until delivery
  Interventions: Other: early management strategy
- Late management GDM group (Experimental): early management of GDM defined as intensive metabolic treatment (diet, physical activity self-blood glucose monitoring according and/or insulin therapy according to the French guidelines). This intensive treatment will begin after the randomization until delivery.
  Interventions: Other: late management strategy

INTERVENTIONS:
Other: late management strategy — late management strategy of GDM defined as no intervention until GDM screening at 24-28 weeks. Between 24-28 weeks gestation, a 75-g OGTT will be done
  Arms: Late management GDM group
Other: early management strategy — early management of GDM defined as intensive metabolic treatment. Intensive treatment involved the following multidisciplinary approach: lifestyle defined by diet and exercise intervention according to the French guidelines
  Arms: Early management GDM group

SUMMARY:
In 2010, the International Association of the Diabetes and Pregnancy Study Groups (IADPSG) panel published consensus-based recommendations on the diagnosis and classification of hyperglycemia in pregnancy. Cognizant that milder degrees of hyperglycemia would also be detected by early pregnancy testing, the IADPSG recommended that fasting plasma glucose (FPG) in the range of 5.1-6.9 mmol/l should be considered diagnostic of early Gestational Diabetes Mellitus (GDM) even if the level of proof for this recommendation is very low regarding to prognosis. This threshold was extrapolated from the FPG value used between 24 and 28 weeks.

In France, a FPG is proposed at the first prenatal visit for women with risk factors of GDM. Early GDM is diagnosed if FPG is ≥ 5.1 mmol/l, leading to an intensive metabolic management. Data have shown that GDM prevalence increased rapidly from 5.9% in 2009 to 9.3% in 2014. 26.9% of women with hyperglycemia during their pregnancy but without known diabetes are treated before 22 weeks' gestation (WG). More recent data from Italy and China, where IADPSG diagnosis criteria were applied, have strongly challenged this recommendation, and showed that early FPG ≥ 5.1mmo/L is poorly predictive of later GDM. No prior studies have demonstrated benefits to early screening and management. In 2016, the IADPSG members have suggested that the use of the FPG threshold ≥5.1 mmol/l for the identification of GDM in early pregnancy is not justified by current evidence

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* Singleton pregnancy
* Early GDM defined by a fasting plasma glucose between 5.1 mmol/l and 6.1 mmol/ with at least one risk factor (age ≥35 years and/or BMI ≥ 25 kg/m2 and/or familial history of diabetes and/or personal history of GDM and/or personal history of macrosomia).
* First prenatal visit prior 20 weeks of gestation at the time of randomization.
* Signed informed consent

Exclusion Criteria:

Diabetic follow-up started at time of inclusion

* Pre-existing diabetes in pregnancy
* Renal impairment
* Hepatic insufficiency
* History of bariatric surgery
* Long time corticosteroids treatment
* Insufficient understanding
* Language difficulties
* Lack of social Insurance
* Person in emergency situation
* Person under the protection of justice (tutelage/ curatorship)
* Persons deprived of their liberty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women with at least one GDM risk factor and a fasting plasma glucose between 5.1 mmol/l and 6.1 mmol/l prior 20 weeks' gestation.
Enrollment: 2010 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The occurrence of materno-fetal complications | at delivery
  Composite endpoint defined by Large for Gestational Age (LGA) (defined by birth weight ≥90th percentile, adjusted for gestational age, sex, maternal BMI, parity, ethnicity) and/or neonatal hypoglycemia and/or shoulder dystocia and/or birth traumatisms

SECONDARY OUTCOMES:
Correlation between composite endpoint (defined in the outcome 1) and the 5 risk factors of GDM | at delivery
  Correlation between composite endpoint (defined in the outcome 1) and the 5 risk factors of GDM (age more or equal to 35 years, BMI more or equal to 25 kg/m2, familial history of diabetes, personal history of GDM, personal history of macrosomia)
Need for insulin during pregnancy | at each 10 days until delivery
  After at least 10 days of dietary and lifestyles measures, if the target are not achieved, women will receive insulin therapy. fastin glucose target <5.1 mmol/ and/or a 2 hour post prandial capillary glucose < 6.6 mmol/l
  at each 10 days a contact with the diabetologist or the nurses for the transmission of the capillary glycaemia either by phone or by the platform 'myDiabby"
Metabolic data: Fasting plasma glucose | at inclusion (because <20 weeks') and an average at 24 28 weeks of gestation
  Change of value of fasting plasma glucose
Metabolic data: HbA1c | at inclusion (because <20 weeks') and an average at 24 28 weeks of gestation
  Change of value of HbA1c
Oral Glucose Tolerance Test (OGTT) | an average at 24 28 weeks of gestation
Percent of GDM women in the late GDM management group according to the IADPSG criteria. | an average at 24 28 weeks of gestation
  IADPSG criteria(fasting glucose more or equal to 5.1 mmol/l and/or 1h more or equal to 10.0 mmol/l and /or 2h more or equal to 8.5 mmol/l
Number of complications in each subgroup of the late GDM management group | at delivery
  Maternal and neonatal complication

CONTACTS AND LOCATIONS:
Overall Officials: Anne VAMBERGUE, Study Director — University Hospital, Lille
Locations (10):
- France (10):
  - CH ARRAS, Arras
  - Hopital Estaing - Chu63 - Clermont Ferrand, Clermont-Ferrand
  - Hop Claude Huriez Chu Lille, Lille
  - Hopital Saint Vincent - Saint Antoine - Lille, Lille
  - Chu Nimes Caremeau - Nimes 9, Nîmes
  - Hopital Haut-Leveque - Chu - Pessac, Pessac
  - Ch Rene Dubos - Pontoise, Pontoise
  - Chu Site Sud (Saint Pierre) - St Pierre, Saint-Pierre
  - Csapa / Hus / Hopital Civil - Strasbourg, Strasbourg
  - Hopital de Rangueil Chu Toulouse, Toulouse